CLINICAL TRIAL: NCT01549782
Title: Effect of a Mixture of Inulin and Fructo-oligosaccharide on Lactobacillus and Bifidobacterium Intestinal Microbiota of Patients Receiving Radiotherapy: a Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Mixture of Prebiotics on Intestinal Microbiota of Patients Receiving Abdominal Radiotherapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Pilar Garci-a Peris, Endocrinologist., Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Prebiotic2005
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Prebiotics; Microbiota; Radiation Therapy Complication; Endometrial Neoplasms
Keywords: Prebiotics; Microbiota; Radiotherapy; Gynaecological Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiber supplement (Active Comparator): 6 gr daily of fibre (50% inulin and 50% FOS). Patients underwent a 1-week run-in period before starting RT and continued taking the same products throughout the treatment course, until three weeks after RT was finished.
  Interventions: Dietary Supplement: Inulin and Fructo-oligosaccharide
- Maltodextrine (Placebo Comparator): 6 gr daily of maltodextrine. Patients underwent a 1-week run-in period before starting RT and continued taking the same products throughout the treatment course, until three weeks after RT was finished.
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Inulin and Fructo-oligosaccharide — 6 gr daily of fibre (50% inulin and 50% FOS). Patients underwent a 1-week run-in period before starting RT and continued taking the same products throughout the treatment course, until three weeks after RT was finished.
  Arms: Fiber supplement
Dietary Supplement: Maltodextrine — 6 gr daily of maltodextrine. Patients underwent a 1-week run-in period before starting RT and continued taking the same products throughout the treatment course, until three weeks after RT was finished.
  Arms: Maltodextrine

SUMMARY:
Abdominal and pelvic radiotherapy (RT) reduces the renewal capacity of the epithelium. Rectal biopsies obtained from patients receiving pelvic RT have revealed atrophy of surface epithelium, acute cryptitis, crypt abscesses, crypt distortion and atrophy, and stromal inflammation. Modifications in intestinal microbiota, such as an increase in the number of pathogens, may contribute to intestinal injury. The prebiotic effect of a carbohydrate is assessed by its capacity to stimulate the proliferation of healthy bacteria (Bifidobacterium, Lactobacillus) rather than pathogenic bacteria (Clostridium, E. coli).

The hypothesis of the study is that a mixture of inulin and fructooligosaccharide could modulate Lactobacillus and Bifidobacterium and reduce the intestinal injury in patients affected of gynaecological cancer and treated with abdominal radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* female gender, age ≥ 18 years, and a diagnosis of gynaecologic cancer requiring postoperative pelvic RT.

Exclusion Criteria:

* previous RT, previous or adjuvant chemotherapy, other types of pelvic tumours or other gynaecologic malignancies, antibiotic or immunosuppressive treatment one week before inclusion or during treatment, and the presence of acute or chronic gastrointestinal disease contraindicating ingestion of the fibre

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes in Lactobacillus and Bifidobacterium populations | 2 months

SECONDARY OUTCOMES:
Changes in calprotectin and DNA levels. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Garcia-Peris, PhD, Principal Investigator — Nutrition Unit. HGU Gregorio Maranon
Locations (1):
- Nutrition Unit. HGU Gregorio Marañón, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Garcia-Peris P, Velasco C, Lozano MA, Moreno Y, Paron L, de la Cuerda C, Breton I, Camblor M, Garcia-Hernandez J, Guarner F, Hernandez M. Effect of a mixture of inulin and fructo-oligosaccharide on Lactobacillus and Bifidobacterium intestinal microbiota of patients receiving radiotherapy: a randomised, double-blind, placebo-controlled trial. Nutr Hosp. 2012 Nov-Dec;27(6):1908-15. doi: 10.3305/nh.2012.27.6.5992. PMID 23588438